CLINICAL TRIAL: NCT00379379
Title: Study of Improving Insulin Sensitivity by Combined Both Electroacupuncture and Drug Therapy
Brief Title: Study of Improving Insulin Sensitivity by Electroacupuncture Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DMR93-IRB-127
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: electroacupuncture, plasma glucose, plasma insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Electroacupuncture

INTERVENTIONS:
Device: electroacupuncture

SUMMARY:
The aim of this study is to find out whether the hypoglycemic and improving insulin resistance effect will appear or not, when EA applying on specific acupoints of NIDDM patients.

DETAILED DESCRIPTION:
Some previous animal model studies reveal that electroacupuncture (EA) applying on specific acupoints, such as Zhongwan and Zusanli acupoint, can reduce plasma glucose levels and encourage insulin secretion, even improve insulin resistance. In this study, we want to observe these results on type II diabetic patients who have been diagnosed in five years under a study design of randomized control trial (RCT) to obtain evidence on clinical.

We undertook a randomized, single blind and sham group controlled study to evaluate the effect of EA with a frequency in 15 Hz and fixed intensity (10 mA) on human Zusanli acupoint. A total of 26 newly diagnostic type II diabetic patients are enrolled in this study. They are randomly divided into 2 groups. There are 13 patients in the experimental group (EG) with EA treatment, and the other 13 patients are divided into control group (CG) with sham treatment. The main outcome is the changes of laboratory parameters between before and 30 minutes after the test.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed NIDDM patient within 5 years
* age between 30 to 65 years old
* controlled BP below 140/90 mmHg
* oral hypoglycemic agent (OHA) therapy with Gliclazide twice per day.

Exclusion Criteria:

* disorders of hemostasis
* patient had received insulin therapy
* severe disease such as CVA, CAD within 6 months
* Arrhythmia history and on pacemaker.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2005-01; Study Completion 2005-12

PRIMARY OUTCOMES:
Hypoglycemic activity, plasma insulin level, HOMA index

SECONDARY OUTCOMES:
Triglyceride, cholesterol, free fatty acid

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Liang Chang, M.D., Ph.D., Principal Investigator — Graduate Institude of Integration Chinese and Western Medicine, China Medical University
Locations (1):
- Graduate Insititude of Integration Chinese And Western Medicine, China Medical University, Taichung, Taiwan

REFERENCES:
- [Background] Chang SL, Lin JG, Chi TC, Liu IM, Cheng JT. An insulin-dependent hypoglycaemia induced by electroacupuncture at the Zhongwan (CV12) acupoint in diabetic rats. Diabetologia. 1999 Feb;42(2):250-5. doi: 10.1007/s001250051146. PMID 10064107
- [Background] Lin JG, Chang SL, Cheng JT. Release of beta-endorphin from adrenal gland to lower plasma glucose by the electroacupuncture at Zhongwan acupoint in rats. Neurosci Lett. 2002 Jun 21;326(1):17-20. doi: 10.1016/s0304-3940(02)00331-2. PMID 12052528
- [Background] Lin JG, Chen WC, Hsieh CL, Tsai CC, Cheng YW, Cheng JT, Chang SL. Multiple sources of endogenous opioid peptide involved in the hypoglycemic response to 15 Hz electroacupuncture at the Zhongwan acupoint in rats. Neurosci Lett. 2004 Aug 5;366(1):39-42. doi: 10.1016/j.neulet.2004.05.003. PMID 15265586
- [Background] Chang SL, Tsai CC, Lin JG, Hsieh CL, Lin RT, Cheng JT. Involvement of serotonin in the hypoglycemic response to 2 Hz electroacupuncture of zusanli acupoint (ST36) in rats. Neurosci Lett. 2005 Apr 29;379(1):69-73. doi: 10.1016/j.neulet.2004.12.057. Epub 2005 Jan 20. PMID 15814202
- [Background] Chang SL, Lin KJ, Lin RT, Hung PH, Lin JG, Cheng JT. Enhanced insulin sensitivity using electroacupuncture on bilateral Zusanli acupoints (ST 36) in rats. Life Sci. 2006 Aug 1;79(10):967-71. doi: 10.1016/j.lfs.2006.05.005. Epub 2006 May 17. PMID 16762373